CLINICAL TRIAL: NCT02213003
Title: Allogeneic Islet Cells Transplanted Onto the Omentum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Diabetes Research Institute Foundation (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140144
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia; Hypoglycemia Unawareness
Keywords: islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islet transplantation (Experimental): Transplantation of at least 5000 islet equivalents/kg of body weight onto the omentum.
  Interventions: Biological: Islet transplantation

INTERVENTIONS:
Biological: Islet transplantation — Transplantation of at least 5000 islet equivalents/kg of body weight onto the Omentum.

SUMMARY:
Current islet transplantation into the portal vein of the liver has shown the unique ability of islets to stabilize blood glucose levels and prevent severe hypoglycemia in a selected group of subjects with Type 1 diabetes. The main limitations of islet transplantation are the need for systemic immunosuppression to maintain function and the loss of islet function over time. Additionally, many studies have demonstrated that the current site of transplantation in the liver is not an ideal site due to several factors. These factors include (1) significant liver inflammation following islet infusion; (2) potential for life-threatening procedure-related complications such as bleeding and thrombosis; (3) high levels of immunosuppressive drugs and GI toxins in the liver contributing to islet toxicity; (4) the inability to retrieve islets after infusion; and (5) development of graft dysfunction in a number of recipients of intrahepatic allogeneic and autologous islets. The implantation of islets into the omentum will allow adequate engraftment of islets onto the omentum and will lead to comparable or superior functional and clinical outcomes than in the traditional intrahepatic site.

DETAILED DESCRIPTION:
Islet transplantation will be performed in subjects with unstable Type 1 diabetes mellitus under permanent immunosuppression. Islets are re-suspended in autologous plasma and distributed on the omental surface by a minimal invasive approach. Cell adherence is achieved by addition of clinical-grade recombinant human thrombin that reacts with plasma to create a biocompatible, degradable gel containing the islet graft. The primary efficacy endpoint is the proportion of subjects with HbA1c ≤6.5% at 1 year AND free of severe hypoglycemic events from Day 28 to Day 365, inclusive, after the islet transplant. The primary safety endpoint is to demonstrate patient safety throughout all stages of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 to 65 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Type1 diabetes with onset of disease at <40 years of age, insulin-dependence for > 5 years at the time of enrollment
5. Absent stimulated c-peptide (<0.3ng/mL) in response to a mixed meal tolerance test.
6. Involvement in intensive diabetes management
7. At least one episode of severe hypoglycemia in the 12 months prior to study enrollment.
8. Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more OR A Hypoglycemia score greater than or equal to the 90th percentile (1047) during the screening period; OR Marked glycemic lability and defined by a lability index score greater than or equal to the 90th percentile (433 mmol/L2/h•wk-1) during the screening period; OR A composite of a Clarke score of 3 or less and a hypoglycemia score greater than or equal to the 75th percentile (423) and a lability index greater than or equal to the 75th percentile (329) during the screening period.
9. Subjects screening data from 20053135 protocol will be accepted for subjects eligible for this study. If 20053135 visit was 12 months prior to enrollment, Visit 2 laboratory should be repeated.

Exclusion Criteria:

1. Body Mass Index (BMI) >30 kg/m2 or patient weight ≤50 kg.
2. Insulin requirement of >1.0 IU/kg/day or <15 U/day.
3. HbA1c >10%.
4. Untreated proliferative diabetic retinopathy.
5. Blood Pressure: SBP >160 mmHg or DBP >100 mmHg.
6. Glomerular filtration rate <80 mL/min/1.73 m2 (calculated).
7. Presence or history of macroalbuminuria (>300mg/g creatinine).
8. Presence or history of panel-reactive anti-HLA antibodies.
9. For female subjects: Serum or urine Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. If sexually active, subject must use at least two medically accepted methods of birth control.
10. Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB).
11. Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
12. Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection within one year prior to study enrollment.
13. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
14. Active alcohol or substance abuse.
15. Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL).
16. A history of Factor V deficiency.
17. Any coagulopathy or medical condition requiring long-term anticoagulant therapy.
18. Severe co-existing cardiac disease,

    1. recent myocardial infarction (within past 6 months)
    2. evidence of ischemia on functional cardiac exam within the last year) left ventricular ejection fraction <30%.
19. Persistent elevation of liver function tests at the time of study entry.
20. Symptomatic cholecystolithiasis.
21. Acute or chronic pancreatitis.
22. Symptomatic peptic ulcer disease.
23. Gastrointestinal disorders potentially interfering with the ability to absorb oral medications.
24. Hyperlipidemia despite medical therapy (fasting LDL cholesterol > 130 mg/dL, fasting triglycerides > 200 mg/dl).
25. Chronic use of systemic steroids, except for the use of ≤5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
26. Treatment with any anti-diabetic medications other than insulin within 4 weeks of enrollment.

23. Use of any investigational agents within 4 weeks of enrollment. 24. Administration of live attenuated vaccine(s) within 2 months of enrollment. 25. Any medical condition that, in the opinion of the investigator, will interfere with the safe participation in the trial.

26. Treatment with any immunosuppressive regimen at the time of enrollment. 27. A previous islet transplant. 28. A previous pancreas transplant 29. Inflammatory bowel disease. 30. History of intestinal obstructions. 31. Previous major abdominal surgery. 32. History of peritonitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
undecided. This is a small phase 1/2 pilot trial.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Islet Transplantation.
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Number of participants with Severe Hypoglycemia in the Past 12 Months and HbA1c < 10% [Count of Participants; unit: Participants] — Number of participants with a Hemoglobin A1c <10 % and at least one episode of severe hypoglycemia in the 12 months prior to study enrollment.
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: A1c </= 6.5% and no Severe Hypoglycemia
Description: Composite outcome measured by the proportion of subjects with HbA1c level of </= 6.5 % and free of severe hypoglycemic events after omentum islet transplant
Time Frame: From day 28 to day 365 after omentum islet transplant
Measure: Number; unit: Proportion of participants
Arm/Group | Islet Transplantation.
Number analyzed (Participants) | 3
Proportion of participants | 0.667

2. Primary Outcome: Procedural Complications
Description: Safety outcome. Post-procedural complications included were: Bleeding, wound infection, hernia, torsion of omentum, gastrointestinal obstruction, abscess, cysts, and need for surgical intervention. Measured by the count of participants with procedural complications.
Time Frame: From day 28 to day 365 after omentum islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: From day 28 to day 365 after omentum islet transplant
Arm/Group | Islet Transplantation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Weight Loss (Metabolism and nutrition disorders) | 2 (2)
Hair Loss (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia/Low Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Left Parotid Glad Inflammation (Gastrointestinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Achilles Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Stress fracture to the non-weight bearing portion of the left calcaneus (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Hypersensitivity reaction to Thymoglobulin (Immune system disorders) | 1 (1)
Macroscopic Hematuria (Renal and urinary disorders) | 1 (1)
Viral Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure-Like Episode (Nervous system disorders) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1)
Laparoscopic removal of displaced intrauterine device and bilateral tubal ligation (Reproductive system and breast disorders) | 1 (1)
Severe Hypoglycemia (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02213003/Prot_SAP_000.pdf